CLINICAL TRIAL: NCT02069249
Title: Sleep, Nutrition and Psychological Functioning in Kindergarten Children: A Longitudinal Intervention Study
Brief Title: Sleep, Nutrition and Psychological Functioning in Kindergarten Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Michal Kahn, PhD student, Laboratory for Children's Sleep-Wake Disorders, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMB-0425-13
Record Dates: First submitted 2014-02-16; First posted 2014-02-24 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Prevention Harmful Effects
Keywords: Preschool children; Sleep problems; Nutrition problems; Online intervention; Psychological functioning
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Nutrition Intervention (Experimental): Healthy Nutrition Intervention (HNI)
  Interventions: Behavioral: Healthy Nutrition intervention
- Healthy Sleep Intervention (Experimental): Healthy Sleep Intervention (HSI)
  Interventions: Behavioral: Healthy Sleep intervention
- Waiting list control (No Intervention): Waiting list control group

INTERVENTIONS:
Behavioral: Healthy Sleep intervention — Healthy Sleep Intervention (HSI)- This online interactive e-learning system will include information for parents on the following topics: (a) establishing appropriate bedtime, including how to assess the sleep needs of their child, how to establish regular bedtime and overall sleep schedule, how to deal with daytime naps; (b) establishing a regular and enjoyable bedtime routine (e.g. bedtime stories); (c) coping with bedtime resistance, setting limits to excessive demands, rewarding appropriate sleep related behaviors; (d) coping with bedtime and nighttime fears, strategies to deal with separation anxieties, fears of darkness, scary imaginative creatures etc; (e) coping with excessive night-wakings and eliminating potential reinforcing consequences; (f) coping with nightmares, night terrors and other parasomnias (e.g., night-walking).
  Arms: Healthy Sleep Intervention
Behavioral: Healthy Nutrition intervention — Healthy Nutrition Intervention (HNI)- This online system will include information for parents on the following issues: (a) increasing awareness and making healthy food choices; (b) increasing appeal of healthy food by games, rewards, and child involvement in preparation and cooking; (c) setting rules regarding proper eating environment, family meals and schedules; (d) limiting the presence of unhealthy food and beverage temptations at home; (e) limiting TV and other screen time and increasing physical activities; (f) encouraging parents to be positive role models for all these principles.
  Arms: Healthy Nutrition Intervention

SUMMARY:
The proposed study has the following aims: (a) to assess the concomitant and longitudinal links between sleep and cognitive, behavioral and emotional functioning in kindergarten children; (b) to assess the immediate and the long-term effects of an intervention to promote healthy sleep habits (HSI) on the child's evolving sleep patterns, as well as on related cognitive, behavioral and health domains; (c) to assess the immediate and the long-term effects of an intervention deigned to promote healthy nutrition (HNI) on the eating habits of children, their weight and BMI measures (the comparison/control group) and (d) to assess the links between eating habits and sleep in kindergarten children.

The main hypotheses of the proposed study are: (a) Shorter and more disrupted sleep would be concomitantly and longitudinally associated with compromised cognitive, emotional and behavioral functioning in kindergarten children; (b) In comparison to the HNI group, children in the HSI group will extend their total sleep time, improve their sleep quality and their sleep schedule will be more stable following the intervention; (c) improvement in sleep habits will be associated with improvement in cognitive, emotional and behavioral functioning; (d) in comparison to the HIS group, children in the HNI group will improve their eating habits, engage in more physical activities and better manage to achieve and maintain an age-appropriate body weight.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children (aged 3-6 years) and their parents

Exclusion Criteria:

* (a) significant health or neurological-developmental problems; (b) severe psychological problems, psychiatric diagnosis or treatment; (c) concurrent psychotherapy or similar interventions; (d) medical sleep problems (e.g., sleep apnea); (e) lack of mastery in Hebrew.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in actigraphic sleep quality (e.g., number of night-wakings, sleep efficiency) and sleep quantity measures | Baseline, 1 week post-intervention
Change in actigraphic sleep quality (e.g., number of night-wakings, sleep efficiency) and sleep quantity measures | Baseline, 6-month follow up
Change in actigraphic sleep quality (e.g., number of night-wakings, sleep efficiency) and sleep quantity measures | 1 week post-intervention, 6 month follow up
Change in parent reported sleep problems (BCSQ) | Baseline, 1 week post-intervention
Change in parent reported sleep problems (BCSQ) | baseline, 6 month follow up
Change in parent reported sleep problems (BCSQ) | 1 week post intervention, 6 month follow up
Change in parent reported child's sleeping and food consumption (derived from Daily sleep and nutrition logs) | Baseline, 1 week post intervention
Change in parent reported child's sleeping and food consumption (derived from Daily sleep and nutrition logs) | Baseline, 6 month follow up
Change in parent reported child's sleeping and food consumption (derived from Daily sleep and nutrition logs) | 1 week post intervention, 6 month follow up
Change in child reported sleep and eating problems | Baseline, 1 week post intervention
Change in child reported sleep and eating problems | Baseline, 6 month follow up
Change in child reported sleep and eating problems | 1 week post intervention, 6 month follow up
Change in parent reported nutrition habits of the child and family | Baseline, 1 week post intervention
Change in parent reported nutrition habits of the child and family | Baseline, 6 month follow up
Change in parent reported nutrition habits of the child and family | 1 week post intervention, 6 month follow up

SECONDARY OUTCOMES:
Change in child psychopathological symptoms (SDQ) | Baseline, 1 week post intervention
Change in child psychopathological symptoms (SDQ) | Baseline, 6 month follow up
Change in child psychopathological symptoms (SDQ) | 1 week post intervention, 6 month follow up
Change in child attention control abilities (computerized tests) | Baseline, 1 week post intervention
Change in child attention control abilities (computerized tests) | Baseline, 6 month follow up
Change in child attention control abilities (computerized tests) | 1 week post intervention, 6 month follow up
Change in child anthropometric measures (height, weight, blood pressure) | Baseline, 1 week post intervention
Change in child anthropometric measures (height, weight, blood pressure) | Baseline, 6 month follow up
Change in child anthropometric measures (height, weight, blood pressure) | 1 week post intervention, 6 month follow up
Change in reported parental Authority (PAQ-R) | Baseline, 1 week post intervention
Change in reported parental Authority (PAQ-R) | Baseline, 6 month follow up
Change in reported parental Authority (PAQ-R) | 1 week post intervention, 6 month follow up
Change in cry tolerance and limit setting abilities | Baseline, 1 week post intervention
Change in cry tolerance and limit setting abilities | Baseline, 6 month follow up
Change in cry tolerance and limit setting abilities | 1 week post intervention, 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Avi Sadeh, Ds.c., Principal Investigator — Tel Aviv University; Geila Rozen, PhD, Principal Investigator — Rambam Health Care Campus; Ron Shaoul, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Tel Aviv University, Tel Aviv, Israel